CLINICAL TRIAL: NCT00324168
Title: Steroids for Corneal Ulcers Trial
Acronym: SCUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas M. Lietman (Other)
Collaborators: Aravind Eye Hospitals, India (Other); Dartmouth-Hitchcock Medical Center (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor-Investigator, Thomas M. Lietman, Prinicpal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H9332-21899-05; U10EY015114-01 (NIH)
Record Dates: First submitted 2006-05-05; First posted 2006-05-10 (Estimated); Results first posted 2013-06-14 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Corneal Ulcer; Eye Infections, Bacterial
Keywords: Bacterial Infections; Eye Diseases; Bacterial Keratitis; Visual Acuity
MeSH Terms: conditions — Corneal Ulcer; Eye Infections, Bacterial; Bacterial Infections; Eye Diseases | interventions — Anti-Bacterial Agents; Moxifloxacin; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Antibiotics; Drug: Topical corticosteroid
- 2 (Placebo Comparator)
  Interventions: Drug: Antibiotics; Drug: Placebo

INTERVENTIONS:
Drug: Antibiotics — moxifloxacin 0.5% every one hour for 48 hours while awake and then every 2 hours until re-epithelialization
  Other Names: Vigamox
Drug: Topical corticosteroid — prednisolone phosphate 1% with preservative four times a day for 1 week, then twice a day for 1 week, and finally once a day for 1 week
  Arms: 1
Drug: Placebo — 0.9% NaCl and preservative (same as in steroid) four times a day for 1 week, then twice a day for 1 week, and finally once a day for 1 week
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether adding topical steroids improves the outcomes of bacterial corneal ulcers, especially visual acuity.

DETAILED DESCRIPTION:
Antimicrobial treatment of a bacterial corneal ulcer is generally effective in eradicating infection. However, "successful" treatment is not always associated with a good visual outcome. The scarring that accompanies the resolution of infection leaves many eyes blind. Some cornea specialists advocate the use of topical corticosteroids along with antibiotics in an effort to reduce immune-mediated tissue damage and scarring. Others fear using steroids to reduce the cornea's immune response will prolong or even exacerbate infection. Ophthalmologists have been divided on this issue for more than 30 years, and both approaches are acceptable according to the American Academy of Ophthalmology's Preferred Practice Patterns. Evidence from animal and human reports is mixed. A single randomized trial saw a non-significant benefit to steroids but was drastically underpowered (20 patients per study arm).

The study is a randomized, double-masked, placebo-controlled trial to determine whether adding topical steroids improves the outcomes of bacterial corneal ulcers. Five hundred bacterial corneal ulcers presenting to the Aravind Eye Hospitals, the University of California, San Francisco (UCSF) Proctor Foundation, and the Dartmouth-Hitchcock Medical Center will be randomized to receive antibiotic plus steroid or antibiotic plus placebo. Participants will be followed closely until re-epithelialization and then rechecked at three weeks, three months and 12 months post enrollment. A subset of patients will be contacted for a follow-up visit four years post enrollment. The primary outcome is best spectacle-corrected visual acuity three months after enrollment, using best spectacle-corrected enrollment visual acuity as a co-variate.

A pilot study was conducted from January 2005 to August 2005 at Aravind Eye Hospital to assess the feasibility and safety and to estimate the sample size of a larger main trial. Forty-two patients with culture-proven bacterial keratitis were enrolled. They were treated and followed up as in the main trial, up to three months from enrollment.

ELIGIBILITY:
Inclusion Criteria

At Presentation:

* Presence of a corneal ulcer at presentation

At Enrollment:

* Presence of bacteria on blood or chocolate agar culture
* Antibiotic given for > 48 hours
* The patient must be able to verbalize a basic understanding of the study after it is explained to the patient, as determined by physician examiner. This understanding must include a commitment to return for f/u visits.
* Appropriate consent

Exclusion Criteria

At Presentation:

* Overlying epithelial defect < 0.75 mm at its greatest width at presentation
* Corneal perforation or impending perforation
* Evidence of fungus on KOH, Giemsa at time of presentation
* Evidence of acanthamoeba by stain
* Evidence of herpetic keratitis by history or exam
* Corneal scar not easily distinguishable from current ulcer
* Use of a topical steroid in the affected eye during the course of the present ulcer, including use after the symptoms of the ulcer started but before presentation
* Use of systemic prednisolone during the course of the present ulcer
* Age less than 16 years (before 16th birthday)
* Bilateral ulcers
* Previous penetrating keratoplasty
* Pregnancy (by history or urine test)
* Immediate steroid use necessary due to surgery or other condition

At Enrollment:

* Evidence of fungus on culture at time of enrollment
* Absence of bacteria on blood or chocolate agar culture
* Best spectacle-corrected vision worse than 6/60 in the fellow eye
* Corneal perforation or descemetocele
* Known allergy to study medications (steroid or preservative)
* No light perception in the affected eye
* Not willing to come to follow-up visits
* Not willing to participate

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-09; Primary Completion 2011-02 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Srinivasan, M.S., O.D., Principal Investigator — Aravind Eye Hospital; Mike Zegans, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center; Nisha Acharya, M.D., M.S., Principal Investigator — Proctor Foundation, UCSF; Thomas M Lietman, M.D., Study Director — Proctor Foundation, UCSF
Locations (5):
- United States (2):
  - Proctor Foundation, UCSF, San Francisco, California
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
- India (3):
  - Aravind Eye Hospital, Coimbatore, Tamil Nadu
  - Aravind Eye Hospital, Madurai, Tamil Nadu
  - Aravind Eye Hospital, Tirunelveli, Tamil Nadu

REFERENCES:
- [Background] Srinivasan M, Mascarenhas J, Rajaraman R, Ravindran M, Lalitha P, Glidden DV, Ray KJ, Hong KC, Oldenburg CE, Lee SM, Zegans ME, McLeod SD, Lietman TM, Acharya NR; Steroids for Corneal Ulcers Trial Group. The steroids for corneal ulcers trial: study design and baseline characteristics. Arch Ophthalmol. 2012 Feb;130(2):151-7. doi: 10.1001/archophthalmol.2011.303. Epub 2011 Oct 10. PMID 21987581
- [Result] Srinivasan M, Mascarenhas J, Rajaraman R, Ravindran M, Lalitha P, Glidden DV, Ray KJ, Hong KC, Oldenburg CE, Lee SM, Zegans ME, McLeod SD, Lietman TM, Acharya NR; Steroids for Corneal Ulcers Trial Group. Corticosteroids for bacterial keratitis: the Steroids for Corneal Ulcers Trial (SCUT). Arch Ophthalmol. 2012 Feb;130(2):143-50. doi: 10.1001/archophthalmol.2011.315. Epub 2011 Oct 10. PMID 21987582
- [Derived] Hammond JH, Hebert WP, Naimie A, Ray K, Van Gelder RD, DiGiandomenico A, Lalitha P, Srinivasan M, Acharya NR, Lietman T, Hogan DA, Zegans ME. Environmentally Endemic Pseudomonas aeruginosa Strains with Mutations in lasR Are Associated with Increased Disease Severity in Corneal Ulcers. mSphere. 2016 Sep 7;1(5):e00140-16. doi: 10.1128/mSphere.00140-16. eCollection 2016 Sep-Oct. PMID 27631025
- [Derived] McClintic SM, Prajna NV, Srinivasan M, Mascarenhas J, Lalitha P, Rajaraman R, Oldenburg CE, O'Brien KS, Ray KJ, Acharya NR, Lietman TM, Keenan JD. Visual outcomes in treated bacterial keratitis: four years of prospective follow-up. Invest Ophthalmol Vis Sci. 2014 May 2;55(5):2935-40. doi: 10.1167/iovs.14-13980. PMID 24618327
- [Derived] Srinivasan M, Mascarenhas J, Rajaraman R, Ravindran M, Lalitha P, Ray KJ, Zegans ME, Acharya NR, Lietman TM, Keenan JD; Steroids for Corneal Ulcers Trial Group. Visual recovery in treated bacterial keratitis. Ophthalmology. 2014 Jun;121(6):1310-1. doi: 10.1016/j.ophtha.2013.12.041. Epub 2014 Mar 5. PMID 24612976
- [Derived] Srinivasan M, Mascarenhas J, Rajaraman R, Ravindran M, Lalitha P, O'Brien KS, Glidden DV, Ray KJ, Oldenburg CE, Zegans ME, Whitcher JP, McLeod SD, Porco TC, Lietman TM, Acharya NR; Steroids for Corneal Ulcers Trial Group. The steroids for corneal ulcers trial (SCUT): secondary 12-month clinical outcomes of a randomized controlled trial. Am J Ophthalmol. 2014 Feb;157(2):327-333.e3. doi: 10.1016/j.ajo.2013.09.025. Epub 2013 Oct 1. PMID 24315294
- [Derived] Oldenburg CE, Lalitha P, Srinivasan M, Manikandan P, Bharathi MJ, Rajaraman R, Ravindran M, Mascarenhas J, Nardone N, Ray KJ, Glidden DV, Acharya NR, Lietman TM. Moxifloxacin susceptibility mediates the relationship between causative organism and clinical outcome in bacterial keratitis. Invest Ophthalmol Vis Sci. 2013 Feb 28;54(2):1522-6. doi: 10.1167/iovs.12-11246. PMID 23385795
- [Derived] Ray KJ, Prajna L, Srinivasan M, Geetha M, Karpagam R, Glidden D, Oldenburg CE, Sun CQ, McLeod SD, Acharya NR, Lietman TM. Fluoroquinolone treatment and susceptibility of isolates from bacterial keratitis. JAMA Ophthalmol. 2013 Mar;131(3):310-3. doi: 10.1001/jamaophthalmol.2013.1718. PMID 23307105
- [Derived] Lalitha P, Srinivasan M, Rajaraman R, Ravindran M, Mascarenhas J, Priya JL, Sy A, Oldenburg CE, Ray KJ, Zegans ME, McLeod SD, Lietman TM, Acharya NR. Nocardia keratitis: clinical course and effect of corticosteroids. Am J Ophthalmol. 2012 Dec;154(6):934-939.e1. doi: 10.1016/j.ajo.2012.06.001. Epub 2012 Sep 5. PMID 22959881
- [Derived] Lalitha P, Srinivasan M, Manikandan P, Bharathi MJ, Rajaraman R, Ravindran M, Cevallos V, Oldenburg CE, Ray KJ, Toutain-Kidd CM, Glidden DV, Zegans ME, McLeod SD, Acharya NR, Lietman TM. Relationship of in vitro susceptibility to moxifloxacin and in vivo clinical outcome in bacterial keratitis. Clin Infect Dis. 2012 May;54(10):1381-7. doi: 10.1093/cid/cis189. Epub 2012 Mar 23. PMID 22447793
- [Derived] Dalmon C, Porco TC, Lietman TM, Prajna NV, Prajna L, Das MR, Kumar JA, Mascarenhas J, Margolis TP, Whitcher JP, Jeng BH, Keenan JD, Chan MF, McLeod SD, Acharya NR. The clinical differentiation of bacterial and fungal keratitis: a photographic survey. Invest Ophthalmol Vis Sci. 2012 Apr 2;53(4):1787-91. doi: 10.1167/iovs.11-8478. PMID 22395880
- [Derived] Sy A, Srinivasan M, Mascarenhas J, Lalitha P, Rajaraman R, Ravindran M, Oldenburg CE, Ray KJ, Glidden D, Zegans ME, McLeod SD, Lietman TM, Acharya NR. Pseudomonas aeruginosa keratitis: outcomes and response to corticosteroid treatment. Invest Ophthalmol Vis Sci. 2012 Jan 25;53(1):267-72. doi: 10.1167/iovs.11-7840. PMID 22159005
- [Derived] Srinivasan M, Lalitha P, Mahalakshmi R, Prajna NV, Mascarenhas J, Chidambaram JD, Lee S, Hong KC, Zegans M, Glidden DV, McLeod S, Whitcher JP, Lietman TM, Acharya NR. Corticosteroids for bacterial corneal ulcers. Br J Ophthalmol. 2009 Feb;93(2):198-202. doi: 10.1136/bjo.2008.147298. Epub 2008 Oct 1. PMID 18829631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 1, 2006 and February 22, 2010, 1,769 patients were screened for the trial and 500 patients were enrolled.
Pre-assignment Details: Common reasons for ineligibility include impending perforation (n=316, 25%), history of a corneal scar in the affected eye (n=123, 10%) and vision worse than 6/60 in the fellow eye (n=119, 9%).
Groups:
- Steroid: Topical corticosteroid : prednisolone phosphate 1% with preservative four times a day for 1 week, then twice a day for 1 week, and finally once a day for 1 week
  Antibiotics : moxifloxacin 0.5% every one hour for 48 hours while awake and then every 2 hours until re-epithelialization
- Placebo: Placebo : 0.9% NaCl and preservative (same as in steroid) four times a day for 1 week, then twice a day for 1 week, and finally once a day for 1 week
  Antibiotics : moxifloxacin 0.5% every one hour for 48 hours while awake and then every 2 hours until re-epithelialization
Period: Overall Study
Arm/Group | Steroid | Placebo
Started | 250 | 250
Completed | 222 | 220
Not Completed | 28 | 30
Not completed — Lost to Follow-up | 19 | 18
Not completed — Death | 3 | 3
Not completed — Patient did not visit in f/u window | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Steroid: Topical corticosteroid : prednisolone phosphate 1% with preservative four times a day for 1 week, BID for 1 week, QD for 1 week
  Antibiotics : moxifloxacin 0.5% every one hour for 48 hours while awake and then every 2 hours until re-epithelialization
- Placebo: Placebo : 0.9% NaCl and preservative (same as in steroid) four times a day for 1 week, BID for 1 week, QD for 1 week
  Antibiotics : moxifloxacin 0.5% every one hour for 48 hours while awake and then every 2 hours until re-epithelialization
- Total: Total of all reporting groups
Arm/Group | Steroid | Placebo | Total
Number analyzed (Participants) | 250 | 250 | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 7
  Between 18 and 65 years | 190 | 198 | 388
  >=65 years | 56 | 49 | 105
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.0 [40.0 to 62.0] | 54.5 [40.0 to 61.0] | 53.0 [40.0 to 61.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 103 | 227
  Male | 126 | 147 | 273
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15
  India | 243 | 242 | 485

OUTCOME MEASURES:

1. Primary Outcome: Best Spectacle-corrected Visual Acuity (BSCVA) in logMAR at 3 Months, Using Best Spectacle-corrected Enrollment Visual Acuity as a Co-variate
Description: LogMAR (logarithm of the Minimum Angle of Resolution) is a measure of visual acuity in which the smaller values indicate better visual acuity.
Time Frame: 3 months from enrollment
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 222 | 220
logMAR | 0.48 [0.42 to 0.53] | 0.49 [0.43 to 0.54]
Statistical Analysis 1: Comparison: Steroid vs Placebo; Test type: Superiority or Other; p = 0.82, Regression, Linear; Adjusted for enrollment BSCVA; Mean Difference (Net) = -0.009, 95% CI 2-sided [-0.085 to 0.068]

2. Secondary Outcome: Infiltrate/Scar Size, Correcting for Infiltrate/Scar Size at Enrollment
Time Frame: 3 months from enrollment
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 222 | 220
mm | 3.07 [2.99 to 3.16] | 3.02 [2.93 to 3.11]
Statistical Analysis 1: Comparison: Steroid vs Placebo; Test type: Superiority or Other; p = 0.40, Regression, Linear; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.09 to 0.15]

3. Secondary Outcome: Best Hard Contact Lens Corrected Visual Acuity Measured in logMAR, Correcting for Best Spectacle Corrected Visual Acuity at Enrollment
Description: as for outcome 1
Time Frame: 3 months from enrollment
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 222 | 220
logMAR | 0.42 [0.36 to 0.47] | 0.41 [0.36 to 0.46]
Statistical Analysis 1: Comparison: Steroid vs Placebo; Test type: Superiority or Other; p = 0.873, Regression, Linear; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.07 to 0.08]

4. Secondary Outcome: Time to Resolution of Epithelial Defect
Description: This outcome measured time from enrollment to resolution of the epithelial defect in days for up to 21 days. For three weeks patients were examined every 3 days for size of epithelial defect until the defect was gone.
Time Frame: From enrollment up to 21 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 222 | 220
days | 9.77 (7.54) [lower limit 7.54] | 9.43 (7.10)
Statistical Analysis 1: Comparison: Steroid vs Placebo; Test type: Superiority or Other; p = 0.44, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.76 to 1.12]

5. Secondary Outcome: Ocular Perforations
Time Frame: At the time of perforation
Measure: Number; unit: participants
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 222 | 220
participants | 7 | 8
Statistical Analysis 1: Comparison: Steroid vs Placebo; Test type: Superiority or Other; p > 0.99, Fisher Exact

6. Secondary Outcome: Best Spectacle-corrected Visual Acuity (BSCVA) in logMAR at 12 Months, Using Best Spectacle-corrected Enrollment Visual Acuity as a Co-variate
Description: as for outcome 1
Time Frame: 12 months from enrollment
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 222 | 220
logMAR | 2.90 [2.80 to 3.01] | 2.87 [2.77 to 2.98]
Statistical Analysis 1: Comparison: Steroid vs Placebo; Test type: Superiority or Other; p = 0.39, Regression, Linear; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.12 to 0.05]

7. Secondary Outcome: Best Spectacle-corrected Visual Acuity (BSCVA) in logMAR Using MIC (Minimum Inhibitory Concentration) to Moxifloxacin as a Covariate
Description: Best spectacle-corrected visual acuity (BSCVA) for this outcome is measured in logMAR (logarithm of the Minimum Angle of Resolution) in which smaller values indicate better visual acuity. Minimum inhibitory concentration (MIC) to moxifloxacin was measured by E test and a log2-transformation of MIC was used in all analyses. In this analysis we add MIC to the model examining BSCVA at 3 months.
Time Frame: 3 months after enrollment
Population: The study population analyzed for this outcome includes only those study subjects for whom an MIC value was available.
Measure: Mean (95% Confidence Interval); unit: logMAR
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 213 | 218
logMAR | 0.50 (0.58) [0.44 to 0.56] | 0.46 (0.49) [0.40 to 0.52]
Statistical Analysis 1: Comparison: Steroid vs Placebo; Test type: Superiority or Other; p = 0.78, Regression, Linear; Mean Difference (Net) = -0.01, 95% CI [-0.09 to 0.07], Standard Error of Mean 0.04

8. Secondary Outcome: Subgroup Analysis Predicting 3 Month Best Spectacle-corrected Visual Acuity (BSCVA) by Causative Organism
Description: BSCVA measured in logMAR will be estimated by causative organism (either Nocardia spp, Streptococcus pneumoniae, Moraxella spp, or Pseudomonas aeruginosa). BSCVA will be examined for each causative organism by mean and standard deviation as well as in a regression model.
Time Frame: 3 months after enrollment
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 222 | 220
logMAR
  Nocardia spp | 0.54 (0.67) | 0.36 (0.64)
  Streptococcus pneumoniae | 0.49 (0.56) | 0.52 (0.53)
  Moraxella spp | 0.46 (0.61) | 0.26 (0.65)
  Pseudomonas aeruginosa | 0.53 (0.54) | 0.45 (0.56)
Statistical Analysis 1: Comparison: Steroid vs Placebo; Nocardia spp; Test type: Superiority or Other; p = 0.30, Regression, Linear; Mean Difference (Net) = 0.12, 95% CI 2-sided [-.011 to 0.35]
Statistical Analysis 2: Comparison: Steroid vs Placebo; Streptococcus pneumoniae; Test type: Superiority or Other; p = 0.86, Regression, Linear; Mean Difference (Net) = -0.01, 95% CI [-0.12 to 0.10]
Statistical Analysis 3: Comparison: Steroid vs Placebo; Moraxella spp; Test type: Superiority or Other; p = 0.65, Regression, Linear; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.34 to 0.55]
Statistical Analysis 4: Comparison: Steroid vs Placebo; Pseudomonas aeruginosa; Test type: Superiority or Other; p = 0.67, Regression, Linear; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.20 to 0.13]

9. Secondary Outcome: Subgroup Analysis Predicting 3 Month Best Spectacle-corrected Visual Acuity (BSCVA) by Visual Acuity Group
Description: Best spectacle-corrected visual acuity (BSCVA) for this subgroup analysis was measured in logMAR and then categorized by equivalent Snellen fractions
Time Frame: 3 months from enrollment
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 222 | 220
logMAR
  <20/40 | 0.06 (0.30) | -0.02 (0.12)
  20/40 to 20/800 | 0.36 (0.43) | 0.38 (0.38)
  Counting fingers (CF) or worse | 1.00 (0.55) | 1.15 (0.61)
Statistical Analysis 1: Comparison: Steroid vs Placebo; <20/40; Test type: Superiority or Other; p = 0.33, Regression, Linear; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.08 to 0.25]
Statistical Analysis 2: Comparison: Steroid vs Placebo; 20/40 to 20/800; Test type: Superiority or Other; p = 0.85, Regression, Linear; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.09 to 0.11]
Statistical Analysis 3: Comparison: Steroid vs Placebo; CF or worse; Test type: Superiority or Other; p = 0.03, Regression, Linear; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.31 to -0.02]

10. Secondary Outcome: Subgroup Analysis of Best Spectacle-corrected Visual Acuity (BSCVA) by Categories of Infiltrate Depth
Description: BSCVA measured in logMAR will be examined by categories infiltrate depth (categorized by depth percentage) by mean and standard deviation as well as in a regression model.
Time Frame: 3 months from enrollment
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 222 | 220
logMAR
  >0-33% | 0.35 (0.50) | 0.26 (0.40)
  >33%-67% | 0.52 (0.57) | 0.47 (0.54)
  >67%-100% | 0.80 (0.61) | 0.86 (0.67)
Statistical Analysis 1: Comparison: Steroid vs Placebo; >0-33%; Test type: Superiority or Other; p = 0.31, Regression, Linear; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.05 to 0.17]
Statistical Analysis 2: Comparison: Steroid vs Placebo; >33%-67%; Test type: Superiority or Other; p = 0.94, Regression, Linear; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.13 to 0.14]
Statistical Analysis 3: Comparison: Steroid vs Placebo; >67%-100%; Test type: Superiority or Other; p = 0.07, Regression, Linear; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.31 to 0.01]

11. Secondary Outcome: Subgroup Analysis Predicting Best Spectacle-corrected Visual Acuity (BSCVA) as Stratified by Categories of Infiltrate/Scar Size
Description: Best-spectacle visual acuity (BSCVA) at 3 months from enrollment is stratified by categories of infiltrate/scar size and examined by treatment arm
Time Frame: 3 months from enrollment
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 222 | 220
logMAR
  0-1.90 mm | 0.18 (0.37) | 0.19 (0.33)
  1.91-2.70 mm | 0.39 (0.51) | 0.29 (0.44)
  2.71-4.06 mm | 0.53 (0.60) | 0.53 (0.53)
  4.07-8.90 mm | 0.85 (0.57) | 0.96 (0.67)
Statistical Analysis 1: Comparison: Steroid vs Placebo; 0-1.90 mm; Test type: Superiority or Other; p = 0.53, Regression, Linear; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.10 to 0.20]
Statistical Analysis 2: Comparison: Steroid vs Placebo; 1.91-2.70 mm; Test type: Superiority or Other; p = 0.95, Regression, Linear; Mean Difference (Net) = 0, 95% CI 2-sided [-0.15 to 0.16]
Statistical Analysis 3: Comparison: Steroid vs Placebo; 2.71-4.06 mm; Test type: Superiority or Other; p = 0.70, Regression, Linear; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.12 to 0.18]
Statistical Analysis 4: Comparison: Steroid vs Placebo; 4.07-8.90 mm; Test type: Superiority or Other; p = 0.07, Regression, Linear; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.31 to 0.01]

ADVERSE EVENTS:
Time Frame: 3 months from enrollment
Arm/Group | Steroid | Placebo
Serious Adverse Events (participants affected / at risk) | 15/250 | 13/250
Other Adverse Events (participants affected / at risk) | 44/250 | 34/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Steroid (N=250) | Placebo (N=250)
Corneal perforation (Eye disorders) | 7 | 8
Death (General disorders) | 7 | 5
Systemic infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Steroid (N=250) | Placebo (N=250)
Increase in hypopyon (Eye disorders) | 4 | 4
Increase in infiltrate size >50% (Eye disorders) | 9 | 4
No healing of epithelial defect by 21 days (Eye disorders) | 44 | 27
Intraocular pressure (IOP) elevated >25mm Hg by <35 mm Hg (Eye disorders) | 2 | 10
Progressive corneal thinning (Eye disorders) | 0 | 2
Other (General disorders) | 9 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No